CLINICAL TRIAL: NCT06833918
Title: The Interplay Between LIPCAR, Cuproptosis, and Α-SMA in the Pathogenesis of Acute Myocardial Infarction and Remodeling
Brief Title: LIPCAR, Cuproptosis, and Α-SMA in the Pathogenesis of AMI and Remodeling
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Shaimaa Ramadan Shakhoun Ata, Dr, Assiut University
Other Study IDs: LIPCAR AMI
Record Dates: First submitted 2025-01-13; First posted 2025-02-19 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-01

CONDITIONS: Acute Myocardial Infarction (AMI)
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples With DNA — Blood Sample Collection For plasma isolation a total of 5 ml of peripheral antecubital venous blood will be obtained in the morning after an overnight fast from each patient within 24 h of the onset of myocardial infarction and from healthy controls in EDTA-containing tubes. The plasma will be separated by centrifugation at 800 g for 10 min. The supernatant plasma samples will be divided into RNase-free Eppendorf tubes and stored at - 80 until analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Genetic: blood sampling — The followings markers will be investigated in plasma samples:
  1. LIPCAR, STAT3 and DDIT3 using quantitative real-time polymerase chain reaction (qRT-PCR)
  2. α-SMA using western blot analysis
  3. Troponin T using ELISA expression
  4. Serum levels of fasting blood glucose (FBG), total cholesterol (TC), triglycerides (TG), and high-density lipoprotein cholesterol (HDL-C), oxidized low-density lipoprotein (ox-LDL) using chemical methods (spectrophotometry). The Friedewald formula was used to compute low-density lipoprotein cholesterol (LDL-C): LDL-Cholesterol =Total cholesterol- (HDL-Cholesterol +Triglycerides/5).

SUMMARY:
The pathophysiology of acute myocardial infarction is multifaceted, involving numerous biological processes. The crosstalk between cuproptosis and remodeling biomarkers may be implicated in the pathogenesis of AMI. Combining cuproptosis, LIPCAR, and α-SMA cardiac recovery analysis may enable more precise identification of diagnostic biomarkers that help for future improvement of treatment and prognosis

DETAILED DESCRIPTION:
Acute myocardial infarction (AMI) is a primary cause of high mortality and disability, which seriously threatens human health across the world (1). AMI is the result of acute interruption of myocardial blood flow followed by myocardial ischemic hypoxic necrosis changes (2). Generally speaking, the traditional risk factors include age, smoking, hypertension, obesity, diabetes, and family history (3). There are two main strategies to reduce the size of myocardial infarction, reduce mortality and improve the prognosis: an early opening of the infarcted vessel and restoration of myocardial blood perfusion, namely known as drug thrombolysis or percutaneous coronary intervention (PCI) surgery (4). Clinically, ECG and high-sensitive cardiac troponins are widely used diagnostic indicators of AMI (5). However, about one-third of patients still do not receive reperfusion therapy as early as possible due to their delayed diagnosis. Therefore, searching for potential biomarkers with high sensitivity and specificity at the beginning of AMI is of great value for individualized diagnosis, early interventional treatment and improvement of prognosis.

The potential use of long noncoding RNAs (LncRNAs) as new biomarkers for cardiovascular diseases is eliciting an increasing interest, because they can be easily detectable and quantifiable in blood samples and are more stable than proteins (6). LncRNAs are a type of transcription products longer than 200 nucleotides that lack protein coding capacity but can epigenetically control both gene expression and protein translation (7). Several lncRNAs were shown to be modulated in the heart or in the circulation in different stress conditions such as AMI and shown to be involved in cardiac remodeling by regulating many biological processes including hypertrophy, fibrosis, autophagy and apoptosis (8). LIPCAR (Long Intergenic noncoding RNA predicting CARdiac remodeling) was identified by Kumarswamy et al. as biomarker of cardiac remodeling" cardiac hypertrophy and fibrosis" and heart failure post-AMI (9). LIPCAR is also a potential biomarker in patients suffering from ST segment elevation myocardial infarction and heart failure post- AMI (10).

Copper is a crucial trace element that plays a role in various pathophysiological processes in the human body. Copper also acts as a transition metal involved in redox reactions, an overabundance of copper is pernicious to the cells, contributing to the generation of reactive oxygen species (ROS). Under prolonged and increased ROS levels, oxidative stress occurs, which has been implicated in different types of regulated cell death (11). The recent discovery of cuproptosis, a copper-dependent regulated cell death pathway that is distinct from other known regulated cell death forms, has raised interest to researchers to reinforce the concept that oxidative stress is a fundamental mechanism of metal-induced toxicity.

The underlying mechanism of copper-induced cell death was unclear until the article "Copper induces cell death by targeting lipoylated TCA cycle proteins" was published by Tsvetkov et al. in 2022. The study sheds light on a novel form of cell death known as cuproptosis, wherein copper binds directly to lipoylated components of the tricarboxylic acid (TCA) cycle, leading to lipoylated protein aggregation and subsequent iron-sulfur cluster protein loss that in turn causes proteotoxic stress and ultimately cell death. The cuproptosis involved in the development of AMI may be dependent on mitochondrial dysfunction (12).

Cuproptosis -related genes (CRGs) were enriched in the regulation of reactive oxygen species metabolic processes, inflammatory response-related pathways, and lipid and atherosclerosis, implying that differential CRGs might participate in the initiation and progression of AMI through these biological processes. Most studies have demonstrated that inflammatory responses play an important role in the initiation and subsequent repair of myocardial infarction (13). Recent studies have linked CRGs: signal transducer and activator of transcription 3 (STAT3), DNA damage-inducible transcript 3 (DDIT3) and AMI, shedding new light on diagnosis and therapy (14, 15). During AMI, the upregulation of DDIT3, a pro-apoptotic transcriptional factor and a feature of endoplasmic reticulum (ER) stress, leads to increased apoptosis of myocardial cells (16). DDIT3 has been shown to have a close relationship with STAT3 in AMI (17).

The α-SMA (alpha-smooth muscle actin) protein plays a crucial role in the regulation of both the proliferation and remodeling of cardiomyocytes, which are the muscle cells of the heart in the first few hours after the onset of coronary occlusion. In the aftermath of a myocardial infarction, it is essential for the damaged heart muscle cells to undergo a process of repair and regeneration to restore normal heart function. Therefore, monitoring and evaluating α-SMA protein expression as a marker of cardiac recovery holds significant importance when assessing the prognosis of patients following acute myocardial infarction (18).

The pathophysiology of acute myocardial infarction is multifaceted, involving numerous biological processes. The crosstalk between cuproptosis and remodeling biomarkers may be implicated in the pathogenesis of AMI. Combining cuproptosis, LIPCAR, and α-SMA cardiac recovery analysis may enable more precise identification of diagnostic biomarkers that help for future improvement of treatment and prognosis.

ELIGIBILITY:
Inclusion Criteria:

* All patients will be subjected to full history taking, meticulous general examination, and local cardiac examination
* Age ≥ 18 years
* AMI diagnosis : clinical, laboratory (troponins level), ECG and coronary angiography indicated occlusion or (≥50% stenosis of any coronary artery or its major branches)

Exclusion Criteria:

* Patients with aortic coarctation,
* Coronary artery bypass grafting surgery,
* Coronary intervention,
* Congestive heart failure,
* Rheumatic heart disease,
* Presence of coronary myocardial bridges,
* Organic cardiac disease such as combined heart valve disease,
* Congenital heart defects,
* Any inflammatory diseases like myocarditis or pericarditis, traumatic cardiac injury or other primary heart diseases,
* Dilated cardiomyopathy,
* Hypertrophic cardiomyopathy,
* Patients complicated with malignant arrhythmias.
* Patients with severe haematological disease,
* Infection as tuberculosis,
* Pulmonary embolism,
* Organ failures or serious lesions (such as brain, lung, liver and kidney),
* Severe autoimmune diseases as arthritis and inflammatory bowel disease,
* Tumours,
* Allergic diseases,
* Connective tissue diseases,
* Trauma,
* And pregnant women or patients with mental disorders such as depression who are unable to cooperate with the study.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The present study will include 50 AMI patients diagnosed and screened based on criteria including persistent chest pain, electrocardiogram changes, and high-sensitivity cardiac troponin I (cTnI) and T testing during their hospital admission to the cardiac catheter unit, department of cardiology, faculty of medicine, Assiut university hospital.
  Patient features will be anonymously analysed in addition to 50 age and gender matched healthy volunteers without history of cardiovascular diseases or other organ issues, no pre-existing or existing cardiovascular symptoms like chest pain during their routine physical examinations in the hospital, normal cardiac enzyme cTnI and T levels, coronary artery stenosis <50% on coronary angiography, and normal ECG parameters as a control group
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
The present study will include two groups: First group: 50 AMI patients and Second group (control): 50 age and gender matched healthy volunteers without history of pre-existing or existing cardiovascular comorbidities with normal cardiac enzymes | 2 years
  The followings markers will be investigated in plasma samples:
  1. LIPCAR, STAT3 and DDIT3 using quantitative real-time polymerase chain reaction (qRT-PCR)
  2. α-SMA using western blot analysis
  3. Troponin T using ELISA expression
  4. Serum levels of fasting blood glucose (FBG), total cholesterol (TC), triglycerides (TG), and high-density lipoprotein cholesterol (HDL-C), oxidized low-density lipoprotein (ox-LDL) using chemical methods (spectrophotometry). The Friedewald formula will be used to compute low-density lipoprotein cholesterol (LDL-C): LDL-Cholesterol =Total cholesterol- (HDL-Cholesterol +Triglycerides/5).
AMI is a myocardial injury event induced by rupture of atherosclerotic plaques and thrombosis. Rapid and accurate identification of AMI in accordance with reducing myocardial cell death has become a critical component for early diagnosis and improvement | 2 years
  The followings markers will be investigated in plasma samples using quantitative real-time polymerase chain reaction (qRT-PCR):
  1. LIPCAR,
  2. STAT3,
  3. DDIT3,
  4. α-SMA and
  5. Troponin T
     * To measure LIPCAR, STAT3 and DDIT3 expression in AMI patients for identifying their role in the pathogenesis of AMI, that could enable further research on its role as a potential therapeutic target.
     * To detect the relationship between LIPCAR, STAT3 and DDIT3 expression and Age, gender, BMI, diabetes mellitus (DM), hypertension (HTN), dyslipidaemia,smoking, and obesity.
     * To detect the relationship between α-SMA protein expression and cardiac regeneration and repair, so that healthcare providers can make more informed decisions regarding treatment strategies, allowing for tailored pharmacological or intervention approaches based on individual patient needs and significantly enhancing heart function and improving the overall quality of life for patients recovering from myocardial infarction.

IPD SHARING:
Plan to Share IPD: Undecided